CLINICAL TRIAL: NCT00071656
Title: Psychosocial Treatment for ADHD Inattentive Type I
Brief Title: Psychosocial Treatment for Attention Deficit Hyperactivity Disorder (ADHD) Type I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: R21MH065927 (NIH); R21MH065927 (NIH); DSIR CT-S
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methods

INTERVENTIONS:
Behavioral: Psychosocial (behavioral) Intervention

SUMMARY:
The purpose of this study is to develop and implement a treatment that focuses on behaviors to reduce symptom severity and functional impairment in patients with Attention Deficit Hyperactivity Disorder, Predominantly Inattentive Type (ADHD-I). The long-term goal of this study is to apply the treatment to larger-scale trials to determine its effectiveness and generalizability.

DETAILED DESCRIPTION:
ADHD-I is a highly prevalent and serious childhood disorder that affects academic and social development. The symptoms of ADHD-I differ from those of the well-studied ADHD Combined Type. Unfortunately, studies of psychosocial interventions for ADHD-I are currently unavailable. Effective treatments for ADHD-I are still needed.

Participants are randomly assigned to receive either a behavioral intervention or treatment as usual for 10 to 12 weeks. The behavioral intervention includes parent and child skill development groups, family meetings, and consultation with the child's teacher to address attention problems and areas of impairment at home and school. Parent and child interviews, teacher and child ratings, and psychoeducational testing are used to assess participants. Participants are assessed post-treatment and at a 2-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* ADHD, Predominantly Inattentive Type
* Public or private school attendance
* English speaking

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60
Dates: Start 2002-09; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- HALP Clinic, Children's Center at Langley Porter, UCSF, San Francisco, California, United States